CLINICAL TRIAL: NCT06043219
Title: The Effects of Action Observation and Motor Imagery on Students' Ability to Locate Anatomical Locations: A Randomised Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Principal Investigator, Paul Chesterton, Professor, Teesside University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: TeessideU23
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Motor Imagery; Action Observation

STUDY DESIGN:
Intervention Model Description: Randomised control trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Groups will be allocated by an academic researcher not involved in the study. The outcome assessor will be blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional Teaching (Active Comparator): Traditional anatomical teaching provided by a powerpoint lecture.
  Interventions: Other: Traditional Teaching
- Action Observational (Experimental): Traditional anatomical teaching via a recorded powerpoint and additionally receiving practice of the task via action observation.
  Interventions: Other: Action Observation; Other: Traditional Teaching
- Action Observational and Motor Imagery (Experimental): Traditional anatomical teaching via a recorded powerpoint and additionally receiving practice of the task via action observation and at the same time imagine themselves executing the same action
  Interventions: Other: Action Observation; Other: Motor Imagery; Other: Traditional Teaching

INTERVENTIONS:
Other: Action Observation — Action observation is defined as watching human movement either via a pre-recorded video or a live demonstration (Eaves et al, 2022). In the current study action observation will be via a pre-recorded video.
  Eaves, D.L., Hodges, N.J., Buckingham, G., Buccino, G. and Vogt, S., 2022. Enhancing motor imagery practice using synchronous action observation. Psychological Research, pp.1-17.
  Arms: Action Observational; Action Observational and Motor Imagery
Other: Motor Imagery — Motor imagery practice is defined as the structured engagement in motor imagery over time for the purpose of acquiring and enhancing motor skills (Eaves et al, 2022).
  Eaves, D.L., Hodges, N.J., Buckingham, G., Buccino, G. and Vogt, S., 2022. Enhancing motor imagery practice using synchronous action observation. Psychological Research, pp.1-17.
  Arms: Action Observational and Motor Imagery
Other: Traditional Teaching — Traditional anatomical teaching via a powerpoint slide deck

SUMMARY:
The aim of this investigation is to measure if additional pedagogical techniques (Action Observation and Motor Imagery) improve student's ability to identify anatomical structures compared to traditional teaching techniques.

DETAILED DESCRIPTION:
The aim of this investigation is to measure if additional pedagogical techniques (Action Observation and Motor Imagery) improve student's ability to identify anatomical structures compared to traditional teaching techniques. Action observation is defined as watching human movement either via a pre-recorded video or a live demonstration. Motor imagery is defined as the mental representation of human movement, including its sensory and motor aspects, without physically executing the action. For example, imagining the feeling and effort of moving your upper-limb to reach out and grasp a glass of water from on top of a table. Motor imagery practice is defined as the structured engagement in motor imagery over time for the purpose of acquiring and enhancing motor skills.

Traditional teaching of anatomy using a common powerpoint based method, will be compared to the traditional powerpoint method plus the addition of action observation techniques or action observation and motor imagery techniques. The investigation, will also look at whether these interventions have an effect on information retention, by retesting the groups at a later date.

ELIGIBILITY:
Inclusion Criteria:

* Level 4 (year one) pre-registration Teesside University physiotherapy/Occupational Therapy/Radiography/Sports Rehab students.
* No previous specific University anatomy training.
* Willing to provide informed consent.

Exclusion Criteria:

* Non Teesside University students
* Healthcare students with previous University level anatomy knowledge (including those with past healthcare degrees).
* Not willing to provide consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Location of key anatomical locations | Immediately post intervention and one week later
  Each participant from each group will be required to required to palpate and locate 4 key anatomical locations from a list of Biceps Femoris Distal Tendon, Tibialis Posterior Tendon, tibiofemoral joint line, Talocrural joint line, Acromioclavicular Joint line, Long Head of Biceps, Glenohumeral joint line. The accuracy of location will be assessed by diagnostic ultrasound.

SECONDARY OUTCOMES:
Vividness of Movement Imagery Questionnaire-2 | Pre- and post intervention (one week later)
  Screening participant ability to conduct motor imagery
Movement Imagery Questionnaire-3 | Pre- and post intervention (one week later)
  Screening participant ability to conduct motor imagery
The Edinburgh Handedness Inventory | Pre intervention
  Screening participants dominant hand

CONTACTS AND LOCATIONS:
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No